CLINICAL TRIAL: NCT02406027
Title: A Randomized, Two-Period, Double-Blind Placebo-Controlled and Open-Label, Multicenter Extension Study to Determine the Long-Term Safety and Tolerability of JNJ-54861911 in Subjects in the Early Alzheimer's Disease Spectrum
Brief Title: An Extension Study to Evaluate the Long-Term Safety and Tolerability of JNJ-54861911 in Participants in the Early Alzheimer's Disease Spectrum
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR106978; 54861911ALZ2004 (Other: Janssen Research & Development, LLC); 2014-004274-41 (EudraCT Number)
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; JNJ-54861911; Placebo
MeSH Terms: conditions — Alzheimer Disease | interventions — atabecestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (5):
- Double-blind Treatment Phase: JNJ-54861911, 10 mg (Experimental): Participants will continue with their current treatment regimen (10 milligram [mg] of JNJ-54861911) established in the parent study of JNJ-54861911. Participants will receive 10 milligram (mg) of JNJ-54861911 orally, once daily from Day 1 up Week 52 in the DB treatment phase.
  Interventions: Drug: JNJ-54861911, 10 mg
- Double-blind Treatment Phase: JNJ-54861911, 25 mg (Experimental): Participants will continue with their current treatment regimen (25 mg of JNJ-54861911) established in the parent study of JNJ-54861911. Participants will receive 25 mg of JNJ-54861911 orally, once daily from Day 1 up Week 52 in the DB treatment phase.
  Interventions: Drug: JNJ-54861911, 25 mg
- Double-blind Treatment Phase: Placebo (Placebo Comparator): Participants will continue with their current treatment regimen established in the parent study of JNJ-54861911. Participants will receive placebo matching to JNJ-54861911 orally, once daily from Day 1 up Week 52 in the DB treatment phase.
  Interventions: Drug: Placebo
- Open-label Phase: JNJ-54861911, 5 mg (Active Comparator): Participants who were receiving JNJ-54861911, 10 mg and placebo in the DB treatment phase, will receive the 5 mg JNJ-54861911 once daily up to end of treatment visit (until registration of JNJ-54861911 or any safety issue) in Open-label phase.
  Interventions: Drug: JNJ-54861911, 10 mg; Drug: JNJ-54861911, 5 mg
- Open-label Phase: JNJ-54861911, 25 mg (Active Comparator): Participants who were receiving JNJ-54861911, 25 mg in the DB treatment phase, will continue to receive the same regimen in open-label treatment phase. Participants who were receiving placebo in the DB treatment phase will be randomly assigned to receive 25 mg of JNJ-54861911 once daily up to end of treatment visit (until registration of JNJ-54861911 or any safety issue) in the open-label treatment phase.
  Interventions: Drug: JNJ-54861911, 25 mg

INTERVENTIONS:
Drug: JNJ-54861911, 10 mg — Participants will self-administer JNJ-54861911 tablet, 10 mg (2*5 mg), orally, once daily.
  Arms: Double-blind Treatment Phase: JNJ-54861911, 10 mg; Open-label Phase: JNJ-54861911, 5 mg
Drug: JNJ-54861911, 25 mg — Participants will self-administer 1 tablet of JNJ-54861911, containing 25 mg orally, once daily.
  Arms: Double-blind Treatment Phase: JNJ-54861911, 25 mg; Open-label Phase: JNJ-54861911, 25 mg
Drug: Placebo — Participants will self administer placebo matching to JNJ-54861911 orally once daily.
  Arms: Double-blind Treatment Phase: Placebo
Drug: JNJ-54861911, 5 mg — Participants will self-administer JNJ-54861911 tablet, 5 mg, orally, once daily.
  Arms: Open-label Phase: JNJ-54861911, 5 mg

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of JNJ-54861911 in participants in the early Alzheimer's disease (AD [progressive brain disease that slowly destroys memory and thinking skills, and eventually even the ability to carry out the simplest tasks]) spectrum that have completed a Phase 1b or Phase 2 clinical trial with JNJ-54861911, who are willing to continue their assigned treatment.

DETAILED DESCRIPTION:
Participants in the early Alzheimer's Disease (AD) spectrum, enrolled in ongoing or future clinical trials with JNJ-54861911 (Phase 1b or Phase 2 studies) will be provided the opportunity to participate in this study upon completion of their treatment period under the parent protocol. The study will consist of a Screening phase and 2 sequential treatment phases (a 12-month double-blind [DB] treatment phase [placebo controlled] and an open-label [OL] phase [active]) followed by an End-of-Treatment visit. Treatment in OL phase will continue until registration of JNJ-54861911; unless safety issues emerge as determined by the Data Review Committee (DRC) that would warrant termination of the study. Blood and cerebrospinal fluid (CSF) samples will be collected to evaluate the plasma and CSF pharmacokinetics of JNJ-54861911, as well as amyloid beta fragments. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the early Alzheimer's disease (AD) spectrum at time of enrollment under the parent protocol and according to its inclusion and exclusion criteria, must have very recently completed their treatment in a Phase 1b or Phase 2 JNJ-54861911 clinical study (example [e.g.], 54861911ALZ2002) under the parent protocol. Enrollment in this study should be completed (Day 1 of double-blind [DB] treatment phase) as soon as possible, but within 6 weeks, following completion of their treatment period under the parent protocol. If not defined under the parent protocol, completion of the treatment period is defined as having completed all study related procedures of the last visit of the treatment period under the parent protocol. A screening phase of up to 12 weeks may be allowed following written approval of the Sponsor
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Each Participants (or their legally acceptable representative and caregiver depending on disease state and local requirements) must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study
* Participants must have a reliable informant (relative, partner, or friend). The informant must be willing to participate as a source of information and has at least weekly contact with the participant (contact can be in-person, via telephone or other audio/visual communication). The informant must have sufficient contact such that the Investigator feels he/she can provide meaningful information about the participant's daily function. If possible, an alternate informant meeting these criteria who can replace the primary informant should be identified prior to randomization

Exclusion Criteria:

* Any condition or situation which, in the opinion of the Investigator, may put the participant at significant risk, may confound the study results, or may interfere significantly with participant's participation in the study
* The use of concomitant medications known to prolong the QT/QTc interval
* Participant has a history of moderate or severe hepatic impairment or severe renal insufficiency unless completely resolved for more than a year. Participant has clinically significant ongoing hepatic, renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, hematologic, rheumatologic, psychiatric or metabolic conditions (e.g., requiring frequent monitoring or medication adjustments or is otherwise unstable)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Chair — Janssen Research & Development, LLC
Locations (17):
- Belgium (2):
  - Ghent
  - Hoboken
- France (3):
  - Montpellier
  - Paris
  - Toulouse
- Germany (5):
  - Essen
  - Homburg
  - Lübeck
  - Tübingen
  - Ulm
- Amsterdam, Netherlands
- Spain (4):
  - Barcelona
  - Madrid
  - Terrasa Barcelona
  - Valencia
- Sweden (2):
  - Mölndal
  - Stockholm

REFERENCES:
- [Derived] Novak G, Streffer JR, Timmers M, Henley D, Brashear HR, Bogert J, Russu A, Janssens L, Tesseur I, Tritsmans L, Van Nueten L, Engelborghs S. Long-term safety and tolerability of atabecestat (JNJ-54861911), an oral BACE1 inhibitor, in early Alzheimer's disease spectrum patients: a randomized, double-blind, placebo-controlled study and a two-period extension study. Alzheimers Res Ther. 2020 May 14;12(1):58. doi: 10.1186/s13195-020-00614-5. PMID 32410694

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed their treatment period as described under the parent protocol in study 54861911ALZ2002 (NCT02260674) or any ongoing/future Phase 1b or Phase 2 atabecestat clinical study were enrolled in this study.
Groups:
- Double-blind Treatment Phase (Period 1): Placebo: Participants received placebo matched to atabecestat orally, once daily from Day 1 up to Week 52 in the Double-blind treatment phase.
- Double-blind Treatment Phase (Period 1): Atabecestat 10 mg: Participants received 10 milligram (mg) of atabecestat orally, once daily from Day 1 up to Week 52 in the Double-blind treatment phase.
- Double-blind Treatment Phase (Period 1): Atabecestat 25 mg: Participants received 25 mg of atabecestat orally, once daily from Day 1 up to Week 52 in the Double-blind treatment phase.
- Open-label (OL) Phase (Period 2): Placebo to Atabecestat 5 mg: Participants who were receiving placebo in the Double-blind treatment phase, received 5 mg atabecestat orally, once daily until registration of atabecestat or any safety issue in Open-label phase.
- OL Phase (Period 2): Placebo to Atabecestat 25 mg: Participants who were receiving placebo in the Double-blind treatment phase, received 25 mg atabecestat orally, once daily until registration of atabecestat or any safety issue in Open-label phase.
- OL Phase (Period 2): Atabecestat 10 mg to Atabecestat 5 mg: Participants who were receiving atabecestat 10 mg in the Double-blind treatment phase, received 5 mg atabecestat orally, once daily until registration of atabecestat or any safety issue in Open-label phase.
- OL Phase (Period 2): Atabecestat 25 mg to Atabecestat 25 mg: Participants who were receiving atabecestat 25 mg in the Double-blind treatment phase continued to receive 25 mg atabecestat orally, once daily until registration of atabecestat or any safety issue in Open-label phase.
Period: Double-blind Treatment Phase (Period 1)
Arm/Group | Double-blind Treatment Phase (Period 1): Placebo | Double-blind Treatment Phase (Period 1): Atabecestat 10 mg | Double-blind Treatment Phase (Period 1): Atabecestat 25 mg | Open-label (OL) Phase (Period 2): Placebo to Atabecestat 5 mg | OL Phase (Period 2): Placebo to Atabecestat 25 mg | OL Phase (Period 2): Atabecestat 10 mg to Atabecestat 5 mg | OL Phase (Period 2): Atabecestat 25 mg to Atabecestat 25 mg
Started | 35 | 29 | 26 | 0 | 0 | 0 | 0
Asymptomatic at Risk | 6 | 8 | 6 | 0 | 0 | 0 | 0
Prodromal | 29 | 21 | 20 | 0 | 0 | 0 | 0
Completed | 29 | 26 | 22 | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 4 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Subject Refused Further Study Treatment | 1 | 0 | 1 | 0 | 0 | 0 | 0
Period: Open-label Phase (Period 2)
Arm/Group | Double-blind Treatment Phase (Period 1): Placebo | Double-blind Treatment Phase (Period 1): Atabecestat 10 mg | Double-blind Treatment Phase (Period 1): Atabecestat 25 mg | Open-label (OL) Phase (Period 2): Placebo to Atabecestat 5 mg | OL Phase (Period 2): Placebo to Atabecestat 25 mg | OL Phase (Period 2): Atabecestat 10 mg to Atabecestat 5 mg | OL Phase (Period 2): Atabecestat 25 mg to Atabecestat 25 mg
Started | 0 | 0 | 0 | 15 | 14 | 26 | 22
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 15 | 14 | 26 | 22
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 4 | 0 | 2
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 11 | 7 | 24 | 19
Not completed — At Spouse Request With PI Agreement | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Subject not Compliant to Study Procedure | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Double-blind safety analysis set included all participants who received study treatment during period 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind Treatment Phase (Period 1): Placebo | Double-blind Treatment Phase (Period 1): Atabecestat 10 mg | Double-blind Treatment Phase (Period 1): Atabecestat 25 mg | Total
Number analyzed (Participants) | 35 | 29 | 26 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (5.15) | 71.4 (7.04) | 67.9 (8.87) | 70 (7.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 12 | 47
  Male | 16 | 13 | 14 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 33 | 25 | 25 | 83
  Unknown or Not Reported | 2 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 35 | 28 | 26 | 89
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Other | 2 | 2 | 1 | 5
  White Non-Hispanic | 33 | 25 | 25 | 83
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 6 | 4 | 3 | 13
  FRANCE | 4 | 2 | 1 | 7
  GERMANY | 4 | 3 | 6 | 13
  NETHERLANDS | 4 | 1 | 3 | 8
  SPAIN | 10 | 17 | 10 | 37
  SWEDEN | 7 | 2 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were events between administration of study drug and up to 3 years that were absent before treatment or that worsened relative to pre-treatment state. An serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 3 years
Population: Safety analysis set included all participants who received at least 1 dose of study drug in the study (during Period 1 and 2).
Measure: Number; unit: Participants
Groups:
- Double-blind Treatment Phase(Period 1): Atabecestat, 25 mg: Participants received 25 mg of atabecestat orally, once daily from Day 1 up to Week 52 in the Double-blind treatment phase.
Arm/Group | Double-blind Treatment Phase (Period 1): Placebo | Double-blind Treatment Phase (Period 1): Atabecestat 10 mg | Double-blind Treatment Phase(Period 1): Atabecestat, 25 mg | Open-label (OL) Phase (Period 2): Placebo to Atabecestat 5 mg | OL Phase (Period 2): Placebo to Atabecestat 25 mg | OL Phase (Period 2): Atabecestat 10 mg to Atabecestat 5 mg | OL Phase (Period 2): Atabecestat 25 mg to Atabecestat 25 mg
Number analyzed (Participants) | 35 | 29 | 26 | 15 | 14 | 26 | 22
Participants
  Number of Participants with TEAEs | 22 | 15 | 21 | 10 | 11 | 19 | 16
  Number of Participants with Serious TEAEs | 3 | 4 | 4 | 2 | 4 | 0 | 1

2. Secondary Outcome: Double-blind Treatment Phase (Period 1): Percent Change From Baseline in Cerebrospinal Fluid (CSF) Amyloid Beta (ABeta) (1-37, 1-38, 1-40, 1-42) Levels
Description: CSF samples were obtained for measuring levels of different ABeta fragments such as ABeta 1-37, ABeta 1-38, ABeta 1-40, and ABeta 1-42. ABeta fragments of different length produced by cleavage of amyloid precursor protein (APP) by beta-secretase (BACE) and gamma-secretase complex in brain and excreted into CSF. Participants were classified as asymptomatic at risk: cognitively and functionally normal (Clinical Dementia Rating Scale score [CDR] =0), but with biomarker pattern consistent with early stage AD (preclinical stage); and prodromal: had some limited cognitive impairment (CDR =0.5), and still functionally normal, with biomarker pattern consistent with early stage (predementia) AD, but had as of yet no dementia (predementia stage). Here, 'Number analyzed=0' signifies that either CSF concentration was below lower limit of quantification for assay or sample was collected under parent study 54861911ALZ2002 (NCT02260674).
Time Frame: Baseline, Double-blind (DB) Day 1 and DB Week 52
Population: The Double-blind (DB) Safety Analysis Set included all participants (asymptomatic at risk and prodromal at baseline) who received study treatment during Period 1. Here 'n' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure at a given time point.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Double-blind Treatment Phase (Period 1): Placebo | Double-blind Treatment Phase (Period 1): Atabecestat 10 mg | Double-blind Treatment Phase(Period 1): Atabecestat, 25 mg
Number analyzed (Participants) | 35 | 29 | 26
Percent change
  CSF ABeta 1-37: Asymptomatic at Risk: DB Day 1: number analyzed (Participants) | 0 | 0 | 0
  CSF ABeta 1-37: Asymptomatic at Risk: DB Week 52: number analyzed (Participants) | 4 | 1 | 1
  CSF ABeta 1-37: Asymptomatic at Risk: DB Week 52 | -9.9 (7.32) | -65.4 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant. | -90.0 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant.
  CSF ABeta 1-37: Prodromal: DB Day 1: number analyzed (Participants) | 3 | 0 | 0
  CSF ABeta 1-37: Prodromal: DB Day 1 | 6.1 (10.09) |  |
  CSF ABeta 1-37: Prodromal: DB Week 52: number analyzed (Participants) | 8 | 8 | 5
  CSF ABeta 1-37: Prodromal: DB Week 52 | -8.8 (17.75) | -62.0 (11.02) | -65.9 (23.16)
  CSF ABeta 1-38: Asymptomatic at Risk: DB Day 1: number analyzed (Participants) | 0 | 0 | 0
  CSF ABeta 1-38: Asymptomatic at Risk: DB Week 52: number analyzed (Participants) | 4 | 3 | 2
  CSF ABeta 1-38: Asymptomatic at Risk: DB Week 52 | -9.3 (7.02) | -42.9 (17.49) | -83.5 (4.84)
  CSF ABeta 1-38: Prodromal: DB Day 1: number analyzed (Participants) | 3 | 0 | 0
  CSF ABeta 1-38: Prodromal: DB Day 1 | 10.2 (15.41) |  |
  CSF ABeta 1-38: Prodromal: DB Week 52: number analyzed (Participants) | 10 | 9 | 10
  CSF ABeta 1-38: Prodromal: DB Week 52 | -9.7 (16.52) | -58.6 (10.21) | -70.4 (23.53)
  CSF ABeta 1-40: Asymptomatic at Risk: DB Day 1: number analyzed (Participants) | 0 | 0 | 0
  CSF ABeta 1-40: Asymptomatic at Risk: DB Week 52: number analyzed (Participants) | 4 | 3 | 2
  CSF ABeta 1-40: Asymptomatic at Risk: DB Week 52 | -9.7 (6.12) | -46.2 (18.22) | -84.6 (5.43)
  CSF ABeta 1-40: Prodromal: DB Day 1: number analyzed (Participants) | 3 | 0 | 0
  CSF ABeta 1-40: Prodromal: DB Day 1 | 8.6 (17.19) |  |
  CSF ABeta 1-40: Prodromal: DB Week 52: number analyzed (Participants) | 12 | 9 | 10
  CSF ABeta 1-40: Prodromal: DB Week 52 | -14.5 (20.48) | -60.7 (13.52) | -72.8 (22.30)
  CSF ABeta 1-42: Asymptomatic at Risk: DB Day 1: number analyzed (Participants) | 0 | 0 | 0
  CSF ABeta 1-42: Asymptomatic at Risk: DB Week 52: number analyzed (Participants) | 4 | 3 | 2
  CSF ABeta 1-42: Asymptomatic at Risk: DB Week 52 | -10.1 (7.81) | -39.6 (24.28) | -76.7 (11.01)
  CSF ABeta 1-42: Prodromal: DB Day 1: number analyzed (Participants) | 3 | 0 | 0
  CSF ABeta 1-42: Prodromal: DB Day 1 | 8.0 (7.44) |  |
  CSF ABeta 1-42: Prodromal: DB Week 52: number analyzed (Participants) | 12 | 9 | 10
  CSF ABeta 1-42: Prodromal: DB Week 52 | -15.0 (20.51) | -52.5 (11.60) | -57.6 (31.42)

3. Secondary Outcome: Double-blind Treatment Phase (Period 1): Percent Change From Baseline in Cerebrospinal Fluid (CSF) Soluble Amyloid Precursor Protein (sAPP) Fragments (sAPP-alpha and sAPP-beta) Levels
Description: The CSF samples were obtained for measuring levels of different soluble amyloid precursor protein (sAPP) fragments (sAPP-alpha, sAPP-beta). Participants were classified as asymptomatic at risk: cognitively and functionally normal (CDR score =0), but with biomarker pattern consistent with early stage alzheimer's disease (AD) (preclinical stage); and prodromal: had some limited cognitive impairment (CDR =0.5), and still functionally normal, with biomarker pattern consistent with early stage (predementia) AD, but had as of yet no dementia (predementia stage). Here, 'Number analyzed=0' signifies that either CSF concentration was below lower limit of quantification for assay or sample was collected under parent study 54861911ALZ2002 (NCT02260674).
Time Frame: Baseline, DB Day 1 and DB Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Double-blind Treatment Phase (Period 1): Placebo | Double-blind Treatment Phase (Period 1): Atabecestat 10 mg | Double-blind Treatment Phase(Period 1): Atabecestat, 25 mg
Number analyzed (Participants) | 35 | 29 | 26
Percent change
  CSF sAPP-alpha: Asymptomatic at Risk: DB Day 1: number analyzed (Participants) | 0 | 0 | 0
  CSF sAPP-alpha: Asymptomatic at Risk: DB Week 52: number analyzed (Participants) | 4 | 3 | 1
  CSF sAPP-alpha: Asymptomatic at Risk: DB Week 52 | -4.7 (12.78) | 50.1 (13.67) | 77.8 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant.
  CSF sAPP-alpha: Prodromal: DB Day 1: number analyzed (Participants) | 3 | 0 | 0
  CSF sAPP-alpha: Prodromal: DB Day 1 | 0.9 (24.97) |  |
  CSF sAPP-alpha: Prodromal: DB Week 52: number analyzed (Participants) | 12 | 9 | 11
  CSF sAPP-alpha: Prodromal: DB Week 52 | -11.2 (14.01) | 60.2 (24.03) | 85.1 (39.35)
  CSF sAPP-Beta: Asymptomatic at Risk: DB Day 1: number analyzed (Participants) | 0 | 0 | 0
  CSF sAPP-Beta: Asymptomatic at Risk: DB Week 52: number analyzed (Participants) | 4 | 3 | 1
  CSF sAPP-Beta: Asymptomatic at Risk: DB Week 52 | -10.8 (8.44) | -57.5 (8.06) | -90.8 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant.
  CSF sAPP-Beta: Prodromal: DB Day 1: number analyzed (Participants) | 3 | 0 | 0
  CSF sAPP-Beta: Prodromal: DB Day 1 | 0.4 (18.93) |  |
  CSF sAPP-Beta: Prodromal: DB Week 52: number analyzed (Participants) | 12 | 9 | 11
  CSF sAPP-Beta: Prodromal: DB Week 52 | -11.7 (14.47) | -63.5 (5.19) | -73.0 (21.79)

4. Secondary Outcome: Double-blind Treatment Phase (Period 1): Percent Change From Baseline in Plasma Amyloid Beta (ABeta) (1-38, 1-40, 1-42) Levels
Description: Plasma samples were obtained for measuring levels of different ABeta fragments such as ABeta 1-38, ABeta 1-40, ABeta 1-42. ABeta fragments of different length were produced by cleavage of APP by beta-secretase (BACE) and gamma-secretase complex in different peripheral tissues, including white blood cells and were measured in plasma. Participants classified as asymptomatic at risk: cognitively and functionally normal (CDR score =0), but with biomarker pattern consistent with early stage AD (preclinical stage); and prodromal: had some limited cognitive impairment (CDR =0.5), and still functionally normal, with biomarker pattern consistent with early stage (predementia) AD, but had as of yet no dementia (predementia stage). Here, 'Number analyzed=0' signifies that either CSF concentration was below lower limit of quantification for assay or sample was collected under parent study 54861911ALZ2002 (NCT02260674).
Time Frame: Baseline, DB Day 1, DB Week 24, and DB Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Double-blind Treatment Phase (Period 1): Placebo | Double-blind Treatment Phase (Period 1): Atabecestat 10 mg | Double-blind Treatment Phase(Period 1): Atabecestat, 25 mg
Number analyzed (Participants) | 35 | 29 | 26
Percent change
  Plasma ABeta 1-38: Asymptomatic at Risk: DB Day 1: number analyzed (Participants) | 0 | 0 | 0
  Plasma ABeta 1-38:Asymptomatic at Risk: DB Week 24: number analyzed (Participants) | 2 | 0 | 0
  Plasma ABeta 1-38:Asymptomatic at Risk: DB Week 24 | -9.9 (0.83) |  |
  Plasma ABeta 1-38: Asymptomatic at Risk:DB Week 52: number analyzed (Participants) | 1 | 0 | 0
  Plasma ABeta 1-38: Asymptomatic at Risk:DB Week 52 | -5.3 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant. |  |
  Plasma ABeta 1-38: Prodromal: DB Day 1: number analyzed (Participants) | 4 | 0 | 3
  Plasma ABeta 1-38: Prodromal: DB Day 1 | -5.0 (10.07) |  | -6.6 (13.56)
  Plasma ABeta 1-38: Prodromal: DB Week 24: number analyzed (Participants) | 4 | 0 | 0
  Plasma ABeta 1-38: Prodromal: DB Week 24 | 3.0 (24.32) |  |
  Plasma ABeta 1-38: Prodromal: DB Week 52: number analyzed (Participants) | 3 | 0 | 0
  Plasma ABeta 1-38: Prodromal: DB Week 52 | 20.3 (35.48) |  |
  Plasma ABeta 1-40: Asymptomatic at Risk: DB Day 1: number analyzed (Participants) | 1 | 1 | 4
  Plasma ABeta 1-40: Asymptomatic at Risk: DB Day 1 | 19.2 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant. | -4.9 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant. | 4.7 (40.27)
  Plasma ABeta 1-40:Asymptomatic at Risk: DB Week 24: number analyzed (Participants) | 5 | 4 | 4
  Plasma ABeta 1-40:Asymptomatic at Risk: DB Week 24 | -2.3 (12.38) | -75.2 (10.16) | -82.6 (5.59)
  Plasma ABeta 1-40:Asymptomatic at Risk: DB Week 52: number analyzed (Participants) | 5 | 4 | 4
  Plasma ABeta 1-40:Asymptomatic at Risk: DB Week 52 | 0.0 (10.85) | -74.9 (6.76) | -80.8 (7.60)
  Plasma ABeta 1-40: Prodromal: DB Day 1: number analyzed (Participants) | 12 | 3 | 7
  Plasma ABeta 1-40: Prodromal: DB Day 1 | 2.9 (15.48) | 25.8 (66.03) | -24.2 (41.31)
  Plasma ABeta 1-40: Prodromal: DB Week 24: number analyzed (Participants) | 21 | 16 | 14
  Plasma ABeta 1-40: Prodromal: DB Week 24 | 8.6 (18.57) | -68.6 (8.20) | -82.5 (7.38)
  Plasma ABeta 1-40: Prodromal: DB Week 52: number analyzed (Participants) | 18 | 15 | 13
  Plasma ABeta 1-40: Prodromal: DB Week 52 | 10.5 (17.09) | -70.9 (9.24) | -75.3 (22.15)
  Plasma ABeta 1-42: Asymptomatic at Risk: DB Day 1: number analyzed (Participants) | 1 | 0 | 0
  Plasma ABeta 1-42: Asymptomatic at Risk: DB Day 1 | -5.9 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant. |  |
  Plasma ABeta 1-42:Asymptomatic at Risk:DB Week 24: number analyzed (Participants) | 3 | 0 | 0
  Plasma ABeta 1-42:Asymptomatic at Risk:DB Week 24 | -7.3 (9.33) |  |
  Plasma ABeta 1-42:Asymptomatic at Risk: DB Week 52: number analyzed (Participants) | 3 | 0 | 0
  Plasma ABeta 1-42:Asymptomatic at Risk: DB Week 52 | -6.0 (2.69) |  |
  Plasma ABeta 1-42: Prodromal: DB Day 1: number analyzed (Participants) | 4 | 0 | 0
  Plasma ABeta 1-42: Prodromal: DB Day 1 | -1.9 (5.54) |  |
  Plasma ABeta 1-42: Prodromal: DB Week 24: number analyzed (Participants) | 8 | 0 | 0
  Plasma ABeta 1-42: Prodromal: DB Week 24 | 15.9 (17.15) |  |
  Plasma ABeta 1-42: Prodromal: DB Week 52: number analyzed (Participants) | 6 | 0 | 0
  Plasma ABeta 1-42: Prodromal: DB Week 52 | 5.1 (17.68) |  |

5. Secondary Outcome: Double-blind Treatment Phase (Period 1): Percent Change From Baseline in Cerebrospinal Fluid (CSF) Tau Protein and Phosphorylated Tau (p-Tau) Protein Level
Description: The CSF samples were obtained for measuring levels of Tau protein and phosphorylated (p)-tau protein. Participants were classified as asymptomatic at risk: cognitively and functionally normal (CDR score =0), but with biomarker pattern consistent with early stage AD (preclinical stage); and prodromal: had some limited cognitive impairment (CDR =0.5), and still functionally normal, with biomarker pattern consistent with early stage (predementia) AD, but had as of yet no dementia (predementia stage). Here, 'Number analyzed=0' signifies that either CSF concentration was below lower limit of quantification for assay or sample was collected under parent study 54861911ALZ2002 (NCT02260674).
Time Frame: Baseline, DB Day 1 and DB Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Double-blind Treatment Phase (Period 1): Placebo | Double-blind Treatment Phase (Period 1): Atabecestat 10 mg | Double-blind Treatment Phase(Period 1): Atabecestat, 25 mg
Number analyzed (Participants) | 35 | 29 | 26
Percent change
  CSF Tau Protein: Asymptomatic at Risk: DB Day 1: number analyzed (Participants) | 0 | 0 | 0
  CSF Tau Protein: Asymptomatic at Risk: DB Week 52: number analyzed (Participants) | 4 | 3 | 1
  CSF Tau Protein: Asymptomatic at Risk: DB Week 52 | -1.4 (14.10) | 3.2 (15.04) | 22.4 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant.
  CSF Tau Protein: Prodromal: DB Day 1: number analyzed (Participants) | 3 | 0 | 0
  CSF Tau Protein: Prodromal: DB Day 1 | 6.1 (6.82) |  |
  CSF Tau Protein: Prodromal: DB Week 52: number analyzed (Participants) | 12 | 9 | 11
  CSF Tau Protein: Prodromal: DB Week 52 | 13.6 (45.55) | 2.1 (13.82) | 1.4 (8.20)
  CSF p-Tau Protein: Asymptomatic at Risk: DB Day 1: number analyzed (Participants) | 0 | 0 | 0
  CSF p-Tau Protein: Asymptomatic at Risk:DB Week 52: number analyzed (Participants) | 4 | 3 | 1
  CSF p-Tau Protein: Asymptomatic at Risk:DB Week 52 | -4.6 (6.47) | -4.9 (1.40) | 8.3 (NA) — Here NA signifies that Standard Deviation could not be calculated for a single participant.
  CSF p-Tau Protein: Prodromal: DB Day 1: number analyzed (Participants) | 3 | 0 | 0
  CSF p-Tau Protein: Prodromal: DB Day 1 | -0.6 (7.81) |  |
  CSF p-Tau Protein: Prodromal: Week 52: number analyzed (Participants) | 12 | 9 | 11
  CSF p-Tau Protein: Prodromal: Week 52 | 2.2 (12.93) | -2.7 (10.52) | -2.6 (8.52)

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Safety analysis set included all participants who received at least 1 dose of study drug in the study (during Period 1 and 2).
Arm/Group | Double-blind Treatment Phase (Period 1): Placebo | Double-blind Treatment Phase (Period 1): Atabecestat 10 mg | Double-blind Treatment Phase (Period 1): Atabecestat 25 mg | Open-label (OL) Phase (Period 2): Placebo to Atabecestat 5 mg | OL Phase (Period 2): Placebo to Atabecestat 25 mg | OL Phase (Period 2): Atabecestat 10 mg to Atabecestat 5 mg | OL Phase (Period 2): Atabecestat 25 mg to Atabecestat 25 mg
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/29 | 0/26 | 0/15 | 0/14 | 0/26 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/35 | 4/29 | 4/26 | 2/15 | 4/14 | 0/26 | 1/22
Other Adverse Events (participants affected / at risk) | 17/35 | 11/29 | 14/26 | 10/15 | 11/14 | 12/26 | 11/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Phase (Period 1): Placebo (N=35) | Double-blind Treatment Phase (Period 1): Atabecestat 10 mg (N=29) | Double-blind Treatment Phase (Period 1): Atabecestat 25 mg (N=26) | Open-label (OL) Phase (Period 2): Placebo to Atabecestat 5 mg (N=15) | OL Phase (Period 2): Placebo to Atabecestat 25 mg (N=14) | OL Phase (Period 2): Atabecestat 10 mg to Atabecestat 5 mg (N=26) | OL Phase (Period 2): Atabecestat 25 mg to Atabecestat 25 mg (N=22)
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Burns Third Degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Transaminases Increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ureteric Obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Treatment Phase (Period 1): Placebo (N=35) | Double-blind Treatment Phase (Period 1): Atabecestat 10 mg (N=29) | Double-blind Treatment Phase (Period 1): Atabecestat 25 mg (N=26) | Open-label (OL) Phase (Period 2): Placebo to Atabecestat 5 mg (N=15) | OL Phase (Period 2): Placebo to Atabecestat 25 mg (N=14) | OL Phase (Period 2): Atabecestat 10 mg to Atabecestat 5 mg (N=26) | OL Phase (Period 2): Atabecestat 25 mg to Atabecestat 25 mg (N=22)
Ear Discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 6 | 0 | 2 | 0 | 0 | 2 | 1
Dry Eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Macular Fibrosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vitreous Floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2 | 1 | 1
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Abscess Neck (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacterial Blepharitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 2 | 1 | 0 | 1 | 0
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 1 | 1
Dermatophytosis of Nail (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 2 | 1 | 3 | 3 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 1 | 0 | 0
Periorbital Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1 | 0 | 3 | 0 | 0
Intraocular Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Transaminases Increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 2 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Complex Regional Pain Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 2 | 3 | 1
Tension Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1
Depressive Symptom (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Nightmare (Psychiatric disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 0
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Nail Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 1
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The major limitation of this study was early termination of the study/program by the sponsor, which resulted in small numbers of participants in groups, precluding meaningful interpretation of some of the analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT02406027/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT02406027/SAP_001.pdf